CLINICAL TRIAL: NCT02457988
Title: COORS: The Cirrhosis Outpatient Optimization, Readmission & Safety Study
Brief Title: The Cirrhosis Outpatient Optimization, Readmission & Safety Study
Acronym: Vivify
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Increased recruitment difficulties
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COORS
Record Dates: First submitted 2015-02-25; First posted 2015-05-29 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2017-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vivify Kit (Experimental): Patients with cirrhosis will undergo home monitoring for 30 days post-discharge through the use of the Vivify kit which contains a wireless tablet with daily medication/diet/symptom questionnaires and vital sign monitoring.
  Interventions: Device: Vivify Kit
- Standard of Care (No Intervention): Patients with cirrhosis will undergo standard of care, which includes a post-discharge lab check and follow-up clinic appointment. Otherwise, no day-to-day monitoring of these patients will occur.

INTERVENTIONS:
Device: Vivify Kit — home telemonitoring devices with vital sign capturing capabilities, i.e. blood pressure, weight, pulse, and specific questionnaires targeted to the cirrhosis diagnosis.
  Arms: Vivify Kit

SUMMARY:
A prospective series comparing care incorporating home monitoring and liver care coordination to conventional care for patients with cirrhosis.

DETAILED DESCRIPTION:
Telemonitoring has been suggested to have potential benefits in patients with cirrhosis. However, to date, no prospective studies exist to support this idea. Hence, the investigators study would like to explore the use of home telemonitoring devices with vital sign capturing capabilities in recently-discharged patients with cirrhosis to decrease 30-day readmissions, mortality and costs.

This is prospective, randomized controlled trial comparing two strategies of post-discharged care in patients with cirrhosis-related hospitalizations.

First treatment arm will incorporate the Vivify home monitoring device into post hospital care.Home monitoring kits include a tablet with wireless internet and vital sign monitoring capabilities (temperature, blood pressure, heart rate, weight and pulse oximetry if needed) and the device has the ability to trigger an alert to the "liver care coordinator."

Second treatment arm will continue the standard of care therapy that all post- hospitalized patients receive upon discharge, i.e. return to clinic appointments, education regarding any signs or worsening symptoms to watch for, as well as contact numbers to connect with their doctor or nurse.

ELIGIBILITY:
Inclusion Criteria:

1. Ascites requiring paracentesis during the hospitalization
2. Hepatic encephalopathy defined as altered mental status that improves after treatment with lactulose
3. Variceal hemorrhage, defined as clinically significant gastrointestinal bleed (tachycardia, hypotension, requirement for blood transfusion, or >2g drop in hemoglobin) and varices seen on endoscopy
4. Spontaneous bacterial peritonitis defined as >250 polymorphonuclear cells per high-power field and/or monomicrobial culture in the ascetic fluid
5. Renal failure in the presence of ascites, defined as a rise in the serum creatinine by 0.5mg/dl (to >1.5mg/dl), with ascites documented on physical exam or ultrasound, or admitted on diuretics for the treatment of ascites
6. Hyponatremia, defined by serum sodium <130 on admission labs
7. Hepatocellular carcinoma as seen on arterial phase MRI or liver biopsy, if tumor is treated and fits within Milan criteria

Exclusion Criteria:

* Admissions for scheduled or elective procedures
* Patients with a comorbid conditions with a life expectancy of less than 12 months or ones that may confound a patient's clinical course

  * Hepatocellular carcinoma
  * Hepatorenal syndrome
  * Hepatopulmonary syndrome
  * Metastatic cancer
  * Chronic kidney disease (pre-dialysis, dialysis)
  * Congestive heart failure
  * Diagnosed dementia
  * HIV/AIDS
  * Pregnancy or planned pregnancy during the study
  * Those managed by palliative care
  * Patients with liver transplants prior to or during the index hospitalization
  * Patients unable to understand study procedures/instructions/use of the home monitoring device
  * Patients unable to stand for <1 minute
  * Patients living in nursing homes or similar institutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of 30-day readmissions between intervention and control group | 30 days
  Compare hospital readmission rates between the intervention group (device) and control group

SECONDARY OUTCOMES:
Number of emergency room visits between the two study groups for ED visits within 30 days post discharge. (composite measure) | 30 days
  Number of ED visits will be measured and compared for both of the groups
Blood pressure control | 30 days
  Overall control of blood pressure between the two groups will be compared
Weight compliance | 30 days
  Weight changes will be monitored and compared between two groups
Medication compliance | 30 days
  Medication compliance will be monitored and compared between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Hommes, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Inflammatory Bowel Diseases, Los Angeles, California, United States

REFERENCES:
- [Background] Volk ML, Tocco RS, Bazick J, Rakoski MO, Lok AS. Hospital readmissions among patients with decompensated cirrhosis. Am J Gastroenterol. 2012 Feb;107(2):247-52. doi: 10.1038/ajg.2011.314. Epub 2011 Sep 20. PMID 21931378
- [Background] Berman K, Tandra S, Forssell K, Vuppalanchi R, Burton JR Jr, Nguyen J, Mullis D, Kwo P, Chalasani N. Incidence and predictors of 30-day readmission among patients hospitalized for advanced liver disease. Clin Gastroenterol Hepatol. 2011 Mar;9(3):254-9. doi: 10.1016/j.cgh.2010.10.035. Epub 2010 Nov 17. PMID 21092762